CLINICAL TRIAL: NCT00117884
Title: A Randomized, Double-blind, Placebo-Controlled, Dose Response Study to Evaluate 851B Gel Delivered Intravaginally Twice a Week for Two, Three-Week Cycles in Women Who Are Positive For High-Risk Genotypes of Human Papillomavirus and Have Mild Cytological Abnormalities
Brief Title: Efficacy of 851B Gel for Treating High-Risk Cervical Human Papillomavirus Infection in Women.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1537-851B; U1111-1127-5850 (Registry Identifier: WHO)
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Papillomavirus Infections
Keywords: Papillomavirus infections;; Cervix Dysplasia
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- 1 (Experimental)
  Interventions: Drug: 851B
- 2 (Experimental)
  Interventions: Drug: 851B
- 3 (Experimental)
  Interventions: Drug: 851B
- 4 (Experimental)
  Interventions: Drug: 851B
- 5 (Experimental)
  Interventions: Drug: 851B
- 6 (Experimental)
  Interventions: Drug: 851B
- 7 (Experimental)
  Interventions: Drug: 851B
- 8 (Experimental)
  Interventions: Drug: 851B
- 9 (Experimental)
  Interventions: Drug: 851B
- 10 (Experimental)
  Interventions: Drug: 851B
- 11 (Experimental)
  Interventions: Drug: 851B

INTERVENTIONS:
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 1
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 2
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 3
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 4
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 5
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 6
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 7
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 8
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 9
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 10
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 11

SUMMARY:
The purpose of this study was to evaluate efficacy of 851B gel over a range of concentrations and dosing regimens on high-risk cervical human papillomavirus infection in women.

DETAILED DESCRIPTION:
Cervical cancer is caused by infection with specific genotypes of the human papillomavirus referred to as oncogenic or high-risk human papillomavirus. Current epidemiologic evidence suggests that 80% of sexually active women will become infected during their lifetime with human papillomavirus and 50% of these infections will be due to high-risk human papillomavirus. With US annual rates of cervical cancer now in the range of 13,000/year, a very substantial number of women are left with uncertainty regarding whether their infection will clear spontaneously or progress to cancer.

Subjects participating in this study were required to visit the clinic for approximately 15 or 16 visits, and maintain a diary of self-dosing and menstruation cycles. The total time of participation in this study was approximately 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be on acceptable method of birth control
* Have a Pap smear result of LSIL or ASCUS
* Is high risk HPV positive

Exclusion Criteria:

* No evidence of high-grade disease or glandular abnormalities,
* Complete visualization of all lesion margins and the transformation zone,
* No uncontrolled significant medical illness or sexually transmitted infections,
* Taking any restricted medications such as interferon, immunomodulators, cytotoxic drugs, investigational drugs, steroids.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Time to clearance of high-risk human papillomavirus infection. | At each visit

SECONDARY OUTCOMES:
Proportion of subjects with evidence of regression to normal cytology. | Screening Visit and Follow-up Visits (Months 6, 8, 14, 20, and 26).
Proportion of subjects with improvement in cervical lesions as rated by the investigator (measured by colposcopy). | At each visit
Proportion of subjects who develop histological evidence of cervical intraepithelial neoplasia. | Visits 1-3 as assigned by group
Time to progression of disease to precancer. | Visits 1-3 as assigned by group
Change in relative light units ratios relative to the positive control from Hybrid Capture 2® assay (semi-quantitatively assessing viral load). | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (23):
- United States (22):
  - Colton, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Boynton Beach, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Savannah, Georgia
  - Louisville, Kentucky
  - Detroit, Michigan
  - Moorestown, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Houston, Texas
  - Renton, Washington
  - Seattle, Washington
  - Spokane, Washington
- Québec, Quebec, Canada